CLINICAL TRIAL: NCT03484975
Title: Novasight Hybrid Intravascular Ultrasound and Optical Coherence Tomography System (IVUS OCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Conavi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EXT-020
Record Dates: First submitted 2018-03-12; First posted 2018-04-02 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Stable Angina; Acute Coronary Syndrome
MeSH Terms: conditions — Angina, Stable; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Observation group (Other): Patients undergoing coronary angiography and intravascular imaging for either diagnostic purposes or for PCI following a presentation with either stable angina or an acute coronary syndrome.
  Interventions: Device: Observation group

INTERVENTIONS:
Device: Observation group — Collect coronary images with a hybrid IVUS OCT system.

SUMMARY:
Collection of coronary images with a hybrid IVUS OCT system.

DETAILED DESCRIPTION:
A prospective observational imaging study in patients undergoing coronary angiography and intravascular imaging for either diagnostic purposes or for PCI following a presentation with either stable angina or an acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old.
2. Patients arriving for coronary angiography or possible PCI with stable angina or acute coronary syndrome (including unstable angina, NSTEMI or STEMI).
3. Patients with STEMI may be undergoing subsequent staged PCI to additional coronary stenoses after the index STEMI event has been successful treated with primary PCI.
4. Vascular access of at least 6F.
5. Patient provides informed, written consent for participation in the study.
6. A target lesion is present in a suitable artery for intravascular imaging.

Exclusion Criteria:

1. Angiographic evidence of severe calcification
2. Marked tortuosity that precludes imaging of a target coronary artery.
3. GFR (Glomerular filtration rate) <35 mL/min.
4. Patients in cardiogenic shock.
5. Women of child bearing potential, in whom pregnancy cannot be excluded.
6. Patients of age < 18 years old.
7. Patients with an allergy to contrast.
8. Patients unable to grant informed, written consent for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Collection of the first human coronary images with the hybrid IVUS OCT technology | Clinical Report Forms (capturing image analysis) will be completed for each case no later then 72 hours after the procedure.
  The hybrid IVUS OCT system permits simultaneous and co-registered acquisition of IVUS and OCT coronary images. IVUS and/or OCT series can be recorded up to 10 cm of the vessel length or up to 20 s of imaging. The physician will review 10 frames and evaluate independently IVUS images, OCT images and the combined IVUS-OCT images for the ability to identify and characterize coronary lesion categories: lipid plaque, calcified plaque, fibrous plaque, thin fibrous cap, positive remodelling and plaque burden. Results, for each frame and imaging modality, of lesion assessment will be tabulated as: a) non-assessable, b) assessable and present, c) assessable and absent. The Clinical Report Form captures tabulated sections for each imaging modality and specific frame selected for lesion evaluation. Results will be presented qualitatively and quantitative as categorical calculations.
  Image interpretation will be performed independently and blinded to clinical and angiographic information.

CONTACTS AND LOCATIONS:
Overall Officials: Tej Sheth, MD, Principal Investigator — Hamilton General Hospital
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided